CLINICAL TRIAL: NCT01218984
Title: A Randomized, Single-Dose Opiate Challenge Study of Medisorb® Naltrexone in Opioid-Using Adults
Brief Title: ALK21-004: Single-dose Opiate Challenge of Medisorb® Naltrexone (VIVITROL®) in Adults Who Use Opioids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Bernard L. Silverman, MD / VP, Clinical Development, Alkermes, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK21-004
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Results first posted 2010-12-13 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Opiate Dependence
Keywords: Opiate Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone; Hydromorphone; Analgesics, Opioid; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Medisorb naltrexone 75 mg (Experimental)
  Interventions: Drug: Medisorb naltrexone 75 mg; Drug: Hydromorphone (10 mg/mL); Drug: Naloxone Challenge and Oral Naltrexone Tolerability Testing
- Medisorb naltrexone 150 mg (Experimental)
  Interventions: Drug: Medisorb naltrexone 150 mg; Drug: Hydromorphone (10 mg/mL); Drug: Naloxone Challenge and Oral Naltrexone Tolerability Testing
- Medisorb naltrexone 300 mg (Experimental)
  Interventions: Drug: Medisorb naltrexone 300 mg; Drug: Hydromorphone (10 mg/mL); Drug: Naloxone Challenge and Oral Naltrexone Tolerability Testing

INTERVENTIONS:
Drug: Medisorb naltrexone 75 mg — Single administration via intramuscular (IM) injection.
  Other Names: Naltrexone for extended-release injectable suspension
  Arms: Medisorb naltrexone 75 mg
Drug: Medisorb naltrexone 150 mg — Single administration via IM injection.
  Other Names: Naltrexone for extended-release injectable suspension
  Arms: Medisorb naltrexone 150 mg
Drug: Medisorb naltrexone 300 mg — Single administration via IM injection.
  Other Names: Naltrexone for extended-release injectable suspension
  Arms: Medisorb naltrexone 300 mg
Drug: Hydromorphone (10 mg/mL) — Increasing doses of 0, 3, 4.5, and 6 mg were administered at baseline (pre-study drug administration). After study drug administration, additional hydromorphone challenge sessions consisting of administering 0, 3, 4.5, and 6 mg were administered at 1-hr intervals at each of the postdose evaluation visits. In addition, at a randomly selected evaluation visit, subjects received four 0 mg (placebo) doses at 1-hour intervals.
  Other Names: Dilaudid-HP®; opioid agonist
Drug: Naloxone Challenge and Oral Naltrexone Tolerability Testing — Administered according to the instructions provided by the respective manufacturer. Testing occurred at least 7 days after the baseline hydromorphone challenge and prior to study drug administration.
  Other Names: Narcan® (naloxone); ReVia® (oral naltrexone)

SUMMARY:
This was a Phase 2, multicenter, randomized, double-blind pilot study in opioid-using adults to assess the presence, duration, and degree of opiate blockade as well as the safety and tolerability of Medisorb® naltrexone (VIVITROL®). Subjects were randomized in a 1:1:1 ratio to receive a single gluteal intramuscular (IM) injection of Medisorb naltrexone 75, 150, or 300 mg.

DETAILED DESCRIPTION:
Potential subjects were screened within 21 days prior to dosing of study drug (Medisorb naltrexone or placebo) on Day 0. Screening evaluations included a baseline hydromorphone challenge session in which increasing doses of hydromorphone (0 mg [placebo], 3 mg, 4.5 mg, and 6 mg) were administered at hourly intervals to produce a cumulative dose-response curve. Throughout the 4-hour challenge period, subject-rated measures (Visual Analog Scale [VAS] questions) and physiological measures (ie, pupil size) were recorded.

As a safety measure, at least 7 days after the baseline hydromorphone challenge, a naloxone challenge was performed followed by a 1-day oral naltrexone tolerability assessment. On Day 0, eligible subjects were administered a single dose of study drug. To assess the level of opiate blockade and surmountability attributable to Medisorb naltrexone, experimental hydromorphone challenge sessions were conducted postdose at Days 7, 14, 21, 28, 42, and 56, with a single placebo hydromorphone challenge administered at a randomly selected visit. Pupil size was measured 15 minutes prior to the first hydromorphone dose and at 15, 30, 45, and minutes after each ascending hydromorphone/placebo for hydromorphone dose. Blood samples for measurement of naltrexone and 6B-naltrexol were obtained at screening and before hydromorphone/placebo administration on Days 7, 14, 21, 28, 42, and 56.

Subjects were monitored for safety through Day 56.

ELIGIBILITY:
Primary Inclusion Criteria:

* Adults who had used opioids: non-medically for at least 1 year; at least once per week for at least some period during their use history; and fewer than 3 times per week on average for the 30 days prior to screening.
* Provided written informed consent
* Demonstrated a positive response to hydromorphone challenge during screening
* Willing to use contraception for study duration if of childbearing potential

Primary Exclusion Criteria:

* Any clinically significant medical condition or laboratory abnormality at screening
* Participated in a clinical trial within prior 30 days
* Dependent on opioids
* Seeking treatment for opioid abuse
* Psychosis or any major mood or anxiety disorder
* Pregnancy or lactation

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-03; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L. Silverman, MD, Study Director — Alkermes, Inc.

REFERENCES:
- [Result] Bigelow GE, Preston KL, Schmittner J, Dong Q, Gastfriend DR. Opioid challenge evaluation of blockade by extended-release naltrexone in opioid-abusing adults: dose-effects and time-course. Drug Alcohol Depend. 2012 Jun 1;123(1-3):57-65. doi: 10.1016/j.drugalcdep.2011.10.018. Epub 2011 Nov 12. PMID 22079773

RESULTS

PARTICIPANT FLOW:
Groups:
- Medisorb Naltrexone 75 mg: Administered as a single gluteal intramuscular (IM) injection
- Medisorb Naltrexone 150 mg; Medisorb Naltrexone 300 mg: Administered as a single gluteal IM injection
Period: Overall Study
Arm/Group | Medisorb Naltrexone 75 mg | Medisorb Naltrexone 150 mg | Medisorb Naltrexone 300 mg
Started | 9 | 8 | 10
Completed | 8 | 6 | 7
Not Completed | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medisorb Naltrexone 75 mg | Medisorb Naltrexone 150 mg | Medisorb Naltrexone 300 mg | Total
Number analyzed (Participants) | 9 | 8 | 10 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 10 | 27
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.22 (9.28) | 42.88 (4.70) | 32.5 (8.02) | 36.48 (8.60)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3
  Male | 8 | 8 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 10 | 27

OUTCOME MEASURES:

1. Primary Outcome: Slope Change From Baseline for Pupil Size
Description: Photographs of subjects' pupils were measured horizontally and vertically, 15 minutes before the first hydromorphone dose and every 15 minutes after each hydromorphone/placebo for hydromorphone dose, for up to 1 hour. Size was the product of vertical and horizontal measures. The slope, determined by linear regression, was used as a summary measure of the dose-response relationship between the hydromorphone dose and pupil size. The steeper the slope, the greater the hydromorphone effect. A slope of zero indicated no evidence of a hydromorphone effect.
Time Frame: 4 weeks (Baseline to Day 28)
Population: Placebo hydromorphone challenge sessions were excluded from the analysis. Results for subjects who discontinued prior to Day 28 were not imputed.
Measure: Mean (Standard Deviation); unit: cm(2)/hr
Arm/Group | Medisorb Naltrexone 75 mg | Medisorb Naltrexone 150 mg | Medisorb Naltrexone 300 mg
Number analyzed (Participants) | 6 | 4 | 6
cm(2)/hr | -0.5540 (0.3473) | -0.3607 (0.3998) | -0.1410 (0.1745)

ADVERSE EVENTS:
Time Frame: 56 Days
Arm/Group | Medisorb Naltrexone 75 mg | Medisorb Naltrexone 150 mg | Medisorb Naltrexone 300 mg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 6/9 | 5/8 | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 75 mg (N=9) | Medisorb Naltrexone 150 mg (N=8) | Medisorb Naltrexone 300 mg (N=10)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Application site rash (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1
Infusion site pain (General disorders) | 1 | 0 | 0
Pain NOS (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury NOS (Injury, poisoning and procedural complications) | 1 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury NOS (Injury, poisoning and procedural complications) | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood in stool (Investigations) | 0 | 0 | 1
Heart rate increased (Investigations) | 1 | 0 | 0
Liver function tests NOS abnormal (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache NOS (Nervous system disorders) | 1 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Factitious disorder NOS (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Dysmennorhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Contusion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritis NOS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Sweating increased (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should a PI wish to disclose results, the Sponsor will review the results communications prior to public release and can embargo results communications for a period of at least 30 days prior to the submission, for review and approval. Revisions will be negotiated in good faith by the Investigator and Sponsor and may be submitted for publication or disclosed by the Investigator only following receipt of written approval from the Sponsor.